CLINICAL TRIAL: NCT03178305
Title: Do Cardiac Health: Advanced New Generation Ecosystem - Phase 2
Acronym: Do CHANGE-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: European Commission (Other); Badalona Serveis Assistencials (Other); Smart Homes (Unknown); ONMI (Unknown); Eindhoven University of Technology (Other); Docobo Ltd. (Industry); Do Something Different (Other); Buddhist Tzu Chi General Hospital (Other); The Industrial Technology Research Institute (Other)
Responsible Party: Principal Investigator, Jos Widdershoven, Prof. Dr., Elisabeth-TweeSteden Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL61660.028.17
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Diseases; Life Style; Quality of Life
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial where patients will be randomly (2:2) assigned to the intervention vs control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Besides the behavior change programme (Do Something Different)
  1. All patients will receive: Fitbit, Beddit, Care-portal, Do CHANGE app (including dietary habits picture taking), CookiT (smart spatula that monitors cooking behavior)
  2. patients with heart failure will, in addition to the above mentioned, be offered a weight scale, blood pressure monitor, and FluiT (smart cup to measure fluid intake).
  3. Patients with hypertension will also be offered a bloodpressure monitor.
  Data from these devices will be gathered and visible for patients (in patient portal) and for their health care provider (health care provider portal). In case of negative results the patient will be contacted by their health care provider (usually the cardiologist).
  Once every week the patients will be contacted to discuss their progress and will be given feedback about their dietary intake.
  Interventions: Behavioral: Do CHANGE
- Care as usual (No Intervention): Patients in this arm will receive care as usual with no restrictions.

INTERVENTIONS:
Behavioral: Do CHANGE — Besides the behavior change programme (Do Something Different)
  1. All patients will receive: Fitbit, Beddit, Care-portal, Do CHANGE app (including dietary habits picture taking), CookiT (smart spatula that monitors cooking behavior)
  2. patients with heart failure will, in addition to the above mentioned, be offered a weight scale, blood pressure monitor, and FluiT (smart cup to measure fluid intake).
  3. Patients with hypertension will also be offered a bloodpressure monitor.
  Data from these devices will be gathered and visible for patients (in patient portal) and for their health care provider (health care provider portal). In case of negative results the patient will be contacted by their health care provider (usually the cardiologist).
  Once every week the patients will be contacted to discuss their progress and will be given feedback about their dietary intake.
  Other Names: Do Something Different
  Arms: Intervention

SUMMARY:
The Do CHANGE service is designed for cardiac patients who could benefit from lifestyle change and a better disease management. The study aims to support patients with behavior change by providing them with devices and behavioral intervention in order to facilitate long-term behavior change.

DETAILED DESCRIPTION:
The focus of the Do CHANGE project is on empowering individuals with high blood pressure, ischemic heart disease or heart failure with tools and services to optimally monitor and manage their real-time health condition and disease. The innovative approach of the Do CHANGE project also involves the patients' surrounding health ecosystem in the process. The traditional difficulties of therapy adherence in a physician-centred care system are radically abandoned and replaced by a patient-centred approach. The approach advocated by Do CHANGE project focuses on the needs of the patient by not only providing them with innovative tools that assess the patient's real-time health condition, but also offer a variety of behavioural alternatives. The main hypothesis of the Do CHANGE project is that patients' disease self-management and lifestyle will improve as compared to self-management of patients who receive the care as usual.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* diagnosed with CAD, HF or HT
* having at least two of the following risk factors: smoking, positive family history, increased cholesterol, diabetes, sedentary lifestyle, psychosocial risk factors.
* Patients should also have access to the Internet and have a smartphone (and sufficient knowledge on using personal computer or smartphone)
* sufficient knowledge of the countries' native language.
* Additional inclusion criteria for HF patients only is to have a previous diagnosis of systolic or diastolic heart failure and experience HF symptoms (e.g. shortness of breath, chest pain, exhaustion).

Exclusion Criteria:

* significant cognitive impairments (e.g. dementia)
* patients who are on the waiting list for heart transplantation
* life expectancy <1 year
* life threatening comorbidities (e.g. cancers),
* a history of psychiatric illness other than anxiety/depression
* patients who do not have access to internet
* patients with insufficient knowledge of the local pilot language (Dutch, Chinese and Catalonian).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Lifestyle | 3 months
  Lifestyle change will be measured with the HPLP-II questionnaire which assesses multiple domains of lifestyle. This will make it possible to compare the two groups.
Quality of Life (QoL) | 3 months
  Quality of life will be assessed with the WHOQoL-Bref which is a validated questionnaire and taps into different domains of quality of life.
Behavioral flexibility | 3 months
  With the Do Something Different purpose designed questionnaire changes in behavioral flexibility will be measured. This programme has previously shown to be effective in changing lifestyle behaviors among physically healthy subjects.

SECONDARY OUTCOMES:
Satisfaction, usability, and acceptance of the intervention | 6 months
  For this purpose the UTAUT-2 questionnaire will be used
Cost effectiveness | 6 months
  the EQ-5D questionnaire will be administered in order to estimate the cost-effectivenss of the intervention.
Health care utilization | 6 months
  Purpose designed questionnaires will be administered to assess health care utilization

OTHER OUTCOMES:
Identification of Subgroups that benefit | 6 months
  Identifying subgroups of patients who are more likely to benefit from this type of approach. Patients with certain demographic and/or psychological profile (Type D personality which will be measured with the DS14 questionnaire) might be more likely to benefit than others.
Effects of intervention on physiological data | 6 months
  Measuring change in patients' physiological data (in the intervention group) in for example, sleep patterns or patients' ECGs, as a result of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jos Widdershoven, MD, PhD, Principal Investigator — Elisabeth-TweeSteden Ziekenhuis
Locations (2):
- Badalona Serveis Assisstencials, Badalona, Barcelona, Spain
- Buddhist Tzu Chi Dalin general hospital, Dalin, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roovers T, Habibovic M, Lodder P, Widdershoven JW, Kop WJ. Changes in heart rate variability during an eHealth behavior change intervention program in patients with cardiovascular disease. Int J Cardiol Heart Vasc. 2024 Nov 22;55:101563. doi: 10.1016/j.ijcha.2024.101563. eCollection 2024 Dec. PMID 39649024
- [Derived] Habibovic M, Piera-Jimenez J, Wetzels M, Widdershoven JWGM, Soedamah-Muthu SS. Associations between behavioral flexibility and health behavior in cardiac patients in the Do CHANGE trials. Health Psychol. 2022 Oct;41(10):710-718. doi: 10.1037/hea0001151. Epub 2022 May 16. PMID 35575702
- [Derived] Piera-Jimenez J, Winters M, Broers E, Valero-Bover D, Habibovic M, Widdershoven JWMG, Folkvord F, Lupianez-Villanueva F. Changing the Health Behavior of Patients With Cardiovascular Disease Through an Electronic Health Intervention in Three Different Countries: Cost-Effectiveness Study in the Do Cardiac Health: Advanced New Generation Ecosystem (Do CHANGE) 2 Randomized Controlled Trial. J Med Internet Res. 2020 Jul 28;22(7):e17351. doi: 10.2196/17351. PMID 32720908
- [Derived] Habibovic M, Gavidia G, Broers E, Wetzels M, Ayoola I, Ribas V, Piera-Jimenez J, Widdershoven J, Denollet J. Type D personality and global positioning system tracked social behavior in patients with cardiovascular disease. Health Psychol. 2020 Aug;39(8):711-720. doi: 10.1037/hea0000823. Epub 2020 Apr 16. PMID 32297772
- [Derived] Broers ER, Widdershoven J, Denollet J, Lodder P, Kop WJ, Wetzels M, Ayoola I, Piera-Jimenez J, Habibovic M; Do CHANGE Consortium. Personalized eHealth Program for Life-style Change: Results From the "Do Cardiac Health Advanced New Generated Ecosystem (Do CHANGE 2)" Randomized Controlled Trial. Psychosom Med. 2020 May;82(4):409-419. doi: 10.1097/PSY.0000000000000802. PMID 32176191
- [Derived] Broers ER, Gavidia G, Wetzels M, Ribas V, Ayoola I, Piera-Jimenez J, Widdershoven JWMG, Habibovic M; Do CHANGE consortium. Usefulness of a Lifestyle Intervention in Patients With Cardiovascular Disease. Am J Cardiol. 2020 Feb 1;125(3):370-375. doi: 10.1016/j.amjcard.2019.10.041. Epub 2019 Nov 6. PMID 31761149
- [Derived] Habibovic M, Broers E, Piera-Jimenez J, Wetzels M, Ayoola I, Denollet J, Widdershoven J. Enhancing Lifestyle Change in Cardiac Patients Through the Do CHANGE System ("Do Cardiac Health: Advanced New Generation Ecosystem"): Randomized Controlled Trial Protocol. JMIR Res Protoc. 2018 Feb 8;7(2):e40. doi: 10.2196/resprot.8406. PMID 29422454